CLINICAL TRIAL: NCT01192152
Title: Bioequivalence Study of the Fixed Dose Combination of 5 mg Saxagliptin/1000 mg Metformin XR (Manufactured in Mt Vernon, IN) Relative to 5 mg of Onglyza and 2 × 500 mg Glucophage XR Coadministered to Healthy Subjects in the Fed State and Steady State Pharmacokinetic Assessment of the Fixed Dose Combination of 5 mg Saxagliptin/1000 mg Metformin XR
Brief Title: Bioequivalence Study of the Fixed Dose Combination of 5 mg Saxagliptin/1000 mg Metformin XR (Manufactured in Mt Vernon, IN) Relative to 5 mg of Onglyza and 2 × 500 mg Glucophage XR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-112
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mg saxagliptin + 2 Glucophage XR 500 mg tablet (Experimental)
  Interventions: Drug: saxagliptin; Drug: Glucophage XR
- FDC tablet (5 mg saxa + 1000 mg metformin XR) (single dose) (Experimental): under fed state, single dose
  Interventions: Drug: saxagliptin + metformin XR (FDC tablet)
- FDC tablet (5 mg saxa + 1000 mg metformin XR) (4 days) (Experimental): under fed state, 4 days
  Interventions: Drug: saxagliptin + metformin XR (FDC tablet)

INTERVENTIONS:
Drug: saxagliptin — Tablets, Oral, 5 mg, once daily, Single dose
  Other Names: Onglyza
  Arms: 5 mg saxagliptin + 2 Glucophage XR 500 mg tablet
Drug: Glucophage XR — Tablets, Oral, 500 mg, once daily, Single dose
  Arms: 5 mg saxagliptin + 2 Glucophage XR 500 mg tablet
Drug: saxagliptin + metformin XR (FDC tablet) — Tablet, Oral, (saxagliptin 5 mg)(metformin XR 1000 mg), once daily, 4 days
  Other Names: Onglyza
  Arms: FDC tablet (5 mg saxa + 1000 mg metformin XR) (4 days); FDC tablet (5 mg saxa + 1000 mg metformin XR) (single dose)

SUMMARY:
The purpose of this study is to demonstrate bioequivalence (BE) of a 5 mg saxagliptin/1000 mg metformin extended release (XR) fixed-dose combination (FDC) tablet (manufactured in Mt Vernon, Indiana) relative to a coadministered 5 mg Onglyza tablet (saxagliptin, manufactured in Mt Vernon, Indiana) and two 500 mg Glucophage XR tablets (metformin XR, manufactured in Evansville, Indiana) in the fed state in healthy subjects.

DETAILED DESCRIPTION:
This study is designed to evaluate if the FDC tablet of 5 mg saxagliptin/1000 mg metformin extended release (manufactured in Mt Vernon, Indiana) is bioequivalent to the coadministered 5 mg saxagliptin tablet plus 2 x 500 mg Glucophage XR tablets (manufactured in Evansville, Indiana)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive
* Ages 18 to 55, inclusive

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Major surgical procedure within 4 weeks prior to randomization
* Positive serology test for HIV, HBV or HCV
* Clinically significant history or presence of any of the following conditions: heart, liver, or kidney disease, neurologic or psychiatric disease
* History of gastrointestinal disease within the past 3 months
* Any clinically significant medical condition that could potentially affect your participation in the study and/or personal well-being, as judged by the investigator
* Donated blood or blood products to a blood bank, blood transfusion or participated in a clinical study (except a screening visit) requiring withdrawal of blood within 4 weeks prior to randomization
* Unable to tolerate oral and/or intravenous (IV) medications
* Unable to tolerate the puncturing of veins for drawing of blood
* Known allergy or hypersensitivity to any component of the study medication
* History of any significant drug allergies (such as anaphylaxis or hepatotoxicity)
* Used any prescription drugs or over the counter products to control acid (for example, Prevacid, Mylanta or Rolaids) within 4 weeks prior to randomization
* Used any other drugs including over the counter medications and herbal preparations within 1 week prior to randomization
* Taken any investigational drug or placebo (inactive drug) within 4 weeks prior to randomization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- [Derived] Boulton DW, Smith CH, Li L, Huang J, Tang A, LaCreta FP. Bioequivalence of saxagliptin/metformin extended-release (XR) fixed-dose combination tablets and single-component saxagliptin and metformin XR tablets in healthy adult subjects. Clin Drug Investig. 2011;31(9):619-30. doi: 10.2165/11590290-000000000-00000. PMID 21819160
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent screening evaluations to determine eligibility within 21 days before dosing, and were admitted to the clinical facility the evening before dosing (Day -1). On Day 1 of Period 1, a total of 30 participants who met all of the inclusion and none of the exclusion criteria were randomly assigned to 1 of 2 treatment sequences.
Groups:
- Treatment Sequence ABC: Treatment A (period 1): 5 mg saxagliptin + 2 Glucophage XR 500 mg under fed conditions; Treatment B (period 2):Fixed dose combination (FDC) tablet (5 mg saxa + 1000 mg metformin XR), single dose, under fed conditions; Treatment C (period 3): FDC tablet (5 mg saxa + 1000 mg metformin XR), once daily for 4 days, under fed conditions. Participants underwent a 2-day washout period between Periods 1 and 2. There was no washout between Periods 2 and 3.
- Treatment Sequence BA: Treatment B (period 1):Fixed dose combination (FDC) tablet (5 mg saxa + 1000 mg metformin XR), single dose, under fed conditions; Treatment A (period 2): 5 mg saxagliptin + 2 Glucophage XR 500 mg under fed conditions. Participants underwent a 2-day washout period between Periods 1 and 2.
Period: Period 1
Arm/Group | Treatment Sequence ABC | Treatment Sequence BA
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — left prematurely (while on treatment B) | 0 | 1
Period: Period 2
Arm/Group | Treatment Sequence ABC | Treatment Sequence BA
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence ABC | Treatment Sequence BA
Started | 15 | 0
Completed | 14 | 0
Not Completed | 1 | 0
Not completed — family emergency | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled and Treated Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 22
  Black or African American | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 17
Height [Mean (Standard Deviation); unit: cm] | 166.85 (9.02)
Weight [Mean (Standard Deviation); unit: kg] | 71.56 (9.39)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.69 (2.70)

OUTCOME MEASURES:

1. Primary Outcome: Saxagliptin Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf])
Time Frame: Periods 1 and 2: pre-dosing, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24, 36 and 48 hours post-dosing.
Population: All treated participants not discontinuing prior to the end of study. One participant in Treatment A was excluded as a result of the inability to estimate with acceptable accuracy a terminal slope for the terminal phase concentration data. Treatment C was administered only during Period 3, and this outcome measure was analyzed for Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Treatment A: Treatment A: 5 mg saxagliptin + 2 Glucophage XR 500 mg tablets, single dose under fed conditions
- Treatment B: Treatment B: Fixed dose combination (FDC) tablet (5 mg saxagliptin + 1000 mg metformin XR), single dose, under fed conditions
- Treatment C: Treatment C: FDC tablet (5 mg saxagliptin + 1000 mg metformin XR), once daily for 4 days, under fed conditions.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ng*hr/mL | 99.45 (18.34) | 105.28 (23.14) |
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; If there was no difference between the bioavailabilities of saxagliptin from the FDC tablet versus saxagliptin from coadministration of a 5-mg saxagliptin tablet plus two 500-mg metformin XR tablets under fed conditions, then 24 subjects would have provided 99% power to conclude bioequivalence (BE) with respect to Cmax and AUC0-inf. If there was a 5% difference, then 24 subjects would have provided 94% and 99% power to conclude BE with respect to Cmax and AUC0-inf; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within 0.800 to 1.250 for both Cmax and AUC0-inf of saxagliptin; Ratio of geometric least squares means = 1.045, 90% CI 2-sided [1.025 to 1.065] — Ratio = Treatment B/Treatment A. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 103.05
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 98.61

2. Secondary Outcome: Saxagliptin Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-t])
Time Frame: as for outcome 1
Population: All treated participants not discontinuing prior to end of study. Treatment C was administered only during Period 3, and this outcome measure was analyzed for Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 0
ng*hr/mL | 97.76 (17.96) | 103.34 (22.73) |
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio of geometric least squares means = 1.035, 90% CI 2-sided [1.009 to 1.062] — Ratio = Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 101.16
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 97.72

3. Secondary Outcome: Saxagliptin Area Under the Plasma Concentration Versus Time Curve From Time 0 to the End of the Dosing Interval (AUC[0-tau])
Description: Dosing interval = 24 hours.
Time Frame: Period 3: pre-dosing on Days 2 and 3; pre-dosing, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, and 24 hours post-dosing on Day 4.
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng*hr/mL |  |  | 19.20 (20.68)

4. Primary Outcome: Saxagliptin Observed Maximum Plasma Concentration (Cmax)
Time Frame: Periods 1 & 2: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24, 36 & 48 hrs post-dosing. Period 3: predosing on Days 2 & 3; predosing, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24 hrs postdosing on Day 4
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
ng/mL | 25.28 (6.40) | 25.75 (6.92) | 25.75 (7.13)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares mean = 0.999, 90% CI 2-sided [0.948 to 1.053] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 24.85
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 24.88

5. Secondary Outcome: Saxagliptin Trough (Predose) Plasma Concentration (Cmin)
Time Frame: Period 3: predosing on Days 2 and 3; predosing, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, and 24 hours postdosing on Day 4.
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng/mL |  |  | 0.28 (0.10)

6. Secondary Outcome: Saxagliptin Average Plasma Concentration Over the Dosing Period (Cavg)
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng/mL |  |  | 4.13 (0.86)

7. Secondary Outcome: Saxagliptin Degree of Fluctuation Over the Dosing Interval (Fluctuation %)
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: percentage of fluctuation
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
percentage of fluctuation |  |  | 611.85 (107.36)

8. Secondary Outcome: Saxagliptin Terminal Half-life (T1/2)
Time Frame: Periods 1 and 2: predosing, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24, 36 and 48 hours postdosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ng*hr/mL | 8.69 (3.71) | 8.85 (4.47) |

9. Secondary Outcome: Saxagliptin Fraction of AUC(0-inf) Contributed by AUC(0-t) (AUC[0-t]/AUC[0-inf])
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ratio | 0.981 (0.010) | 0.982 (0.008) |

10. Secondary Outcome: Saxagliptin Time to Achieve the Observed Maximum Plasma Concentration (Tmax)
Time Frame: Periods 1 & 2:predose, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24, 36, 48 hours postdose. Period 3: predose on Days 2 & 3; predose, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24 hours postdose on Day 4.
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
hour | 1.88 (0.87) | 1.51 (0.64) | 1.35 (0.51)

11. Secondary Outcome: 5-hydroxy Saxagliptin AUC(0-inf)
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ng*hr/mL | 298.80 (69.32) | 296.99 (69.35) |

12. Secondary Outcome: 5-hydroxy Saxagliptin AUC(0-t)
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 0
ng*hr/mL | 293.06 (68.28) | 289.37 (68.72) |

13. Secondary Outcome: 5-hydroxy Saxagliptin AUC(0-tau)
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng*hr/mL |  |  | 318.47 (54.95)

14. Secondary Outcome: 5-hydroxy Saxagliptin Cmax
Time Frame: as for outcome 10
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
ng/mL | 54.69 (17.00) | 51.32 (16.19) | 59.87 (13.83)

15. Secondary Outcome: 5-hydroxy Saxagliptin Cmin
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng/mL |  |  | 1.51 (0.22)

16. Secondary Outcome: 5-hydroxy Saxagliptin Cavg
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng/mL |  |  | 13.27 (2.29)

17. Secondary Outcome: 5-hydroxy Saxagliptin Fluctuation %
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: percentage of fluctuation
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
percentage of fluctuation |  |  | 437.09 (43.97)

18. Secondary Outcome: 5-hydroxy Saxagliptin T1/2
Time Frame: Periods 1 and 2: predosing, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 18, 24, 36 and 48 hours post-dosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ng*hr/mL | 13.48 (1.78) | 13.82 (2.52) |

19. Secondary Outcome: 5-hydroxy Saxagliptin AUC(0-t)/AUC(0-inf)
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ratio | 0.975 (0.009) | 0.973 (0.010) |

20. Secondary Outcome: 5-hydroxy Saxagliptin Tmax
Time Frame: as for outcome 10
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
hour | 2.69 (0.80) | 2.27 (0.84) | 2.05 (0.57)

21. Primary Outcome: Metformin AUC(0-inf)
Time Frame: as for outcome 8
Population: All treated participants not discontinuing prior to end of study. 2 participants in Treatment A & 1 in Treatment B were excluded due to the inability to estimate with acceptable accuracy a terminal slope for terminal phase concentration data. Treatment C administered only during Period 3, and this outcome measure was analyzed for Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 27 | 29 | 0
ng*hr/mL | 10336.18 (3066.13) | 9211.29 (3364.24) |
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; If there was no difference between the bioavailabilities of metformin from the FDC tablet versus metformin from coadministration of a 5-mg saxagliptin tablet plus two 500-mg metformin XR tablets under fed conditions, then 24 subjects would have provided 99% power to conclude BE with respect to Cmax and AUC0-inf. If there was a 5% difference, then 24 subjects would have provided at least 99% power to conclude BE with respect to Cmax and AUC0-inf; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios of geometric means were entirely contained within 0.800 to 1.250 for both Cmax and AUC0-inf of metformin; ratio of geometric least squares means = 0.894, 90% CI 2-sided [0.833 to 0.959] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Treatment B; Geometric least squares mean for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 8713.4
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares mean for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 9746.3

22. Secondary Outcome: Metformin AUC(0-t)
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 0
ng*hr/mL | 9734.38 (3123.76) | 8846.36 (3304.75) |
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; ratio of geometric least squares means = 0.906, 90% CI 2-sided [0.848 to 0.968] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 8377.8
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares mean for Treatment A; Test type: Superiority or Other; Geometric least squares mean (ng*hr/mL) = 9246.8

23. Secondary Outcome: Metformin AUC(0-tau)
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng*hr/mL |  |  | 9501.81 (4001.00)

24. Primary Outcome: Metformin Cmax
Time Frame: as for outcome 10
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
ng/mL | 1184.07 (276.12) | 1078.67 (221.72) | 979.93 (267.58)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 21, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ratio of geometric least squares means = 0.917, 90% CI 2-sided [0.859 to 0.980] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 1055.9
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 1151.2

25. Secondary Outcome: Metformin Cmin
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng/mL |  |  | 105.04 (88.09)

26. Secondary Outcome: Metformin Cavg
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
ng/mL |  |  | 395.91 (166.71)

27. Secondary Outcome: Metformin Fluctuation %
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: percentage of fluctuation
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 14
percentage of fluctuation |  |  | 240.06 (73.54)

28. Secondary Outcome: Metformin T1/2
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 28 | 30 | 0
ng*hr/mL | 13.02 (6.15) | 12.94 (6.74) |

29. Secondary Outcome: Metformin AUC(0-inf) Contributed by AUC(0-t)(AUC[0-t]/AUC[0-inf])
Time Frame: as for outcome 8
Population: All treated participants not discontinuing prior to end of study. 2 participants in Treatment A & 1 in Treatment B were excluded as a result of the inability to estimate with acceptable accuracy a terminal slope for terminal phase concentration data. Treatment C was administered only during Period 3, & this measure was analyzed for Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 27 | 29 | 0
ratio | 0.967 (0.029) | 0.963 (0.034) |

30. Secondary Outcome: Metformin Tmax
Time Frame: as for outcome 10
Population: All treated participants not discontinuing prior to end of study.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
hour | 4.38 (0.73) | 4.84 (0.91) | 5.00 (1.30)

31. Secondary Outcome: Safety: Adverse Events (AEs), Discontinuations Due to AEs, Deaths, and Serious AEs (SAEs)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: AEs: from initiation of study drug administration on morning of Day 1/Period 1 through study discharge. SAEs: from date of written consent until 30 days after discontinuation of dosing or participation in study if last scheduled visit occurred later.
Population: All subjects who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
participants
  Number of Participants With At Least 1 AE | 3 | 3 | 4
  Discontinuation Due to AE | 0 | 0 | 0
  Deaths | 0 | 0 | 0
  SAEs | 0 | 0 | 0

32. Secondary Outcome: Safety: Clinically Significant Laboratory, Vital Sign, Physical Examination, and/or 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Abnormalities considered clinically significant and/or reported as an AE by the investigator.
Time Frame: From Day 1 of Period 1 to Day 3 of Period 2 for participants in Treatment Sequence BA and Day 5 of Period 3 for participants in Treatment Sequence ABC
Population: All subjects who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 30 | 14
participants
  Clinical Laboratory Abnormalities | 0 | 0 | 0
  Vital Sign Abnormalities | 0 | 0 | 0
  Physical Examination Abnormalities | 0 | 0 | 1
  12-Lead ECG Abnormalities | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Saxa 5mg + 2x500mg Metformin, Fed: 5 mg saxagliptin + 2 Glucophage XR 500 mg tablets, single dose under fed conditions
- Saxa 5mg/1000mg Metformin, Fed: Fixed dose combination (FDC) tablet (5 mg saxagliptin + 1000 mg metformin XR), single dose, under fed conditions
- Saxa 5mg/500mg Metformin, Fed 4 Days: FDC tablet (5 mg saxagliptin + 1000 mg metformin XR), once daily for 4 days, under fed conditions.
Arm/Group | Saxa 5mg + 2x500mg Metformin, Fed | Saxa 5mg/1000mg Metformin, Fed | Saxa 5mg/500mg Metformin, Fed 4 Days
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/14
Other Adverse Events (participants affected / at risk) | 3/29 | 3/30 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxa 5mg + 2x500mg Metformin, Fed (N=29) | Saxa 5mg/1000mg Metformin, Fed (N=30) | Saxa 5mg/500mg Metformin, Fed 4 Days (N=14)
HEADACHE (Nervous system disorders) | 0 | 2 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 2
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 0 | 1
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.